CLINICAL TRIAL: NCT05628623
Title: Eradicating Measurable Residual Disease in Patients With Acute Myeloid Leukemia (AML) Prior to StEm Cell Transplantation (ERASE): A MyeloMATCH Treatment Trial
Brief Title: Testing the Use of Combination Therapy in Patients With Persistent Low Level Acute Myeloid Leukemia (AML) Following Initial Treatment
Acronym: ERASE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM2YA-EA01
Record Dates: First submitted 2022-11-18; First posted 2022-11-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; venetoclax; CPX-351; Daunorubicin; Azacitidine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 1 of 4 arms in a 1:1:1:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A: Cytarabine (Active Comparator): Patients will participate for 2 cycles. Each cycle is 28 days.
  For Core Binding Factor (CBF) leukemia patients: Cytarabine 3000 mg/m2 IV twice daily (BID), 12 hours apart x 6 doses either on Days 1, 3, and 5 OR Days 1, 2, and 3 (per institutional preference)
  For non-Core Binding Factor (CBF) leukemia patients: Cytarabine 1500 mg/m2 IV twice daily (BID), 12 hours apart x 6 either on Days 1, 3, and 5 OR Days 1, 2, and 3 (per institutional preference)
  Interventions: Drug: Cytarabine
- Arm B: Cytarabine + Venetoclax (Experimental): Patients will participate for 2 cycles. Each cycle is 28 days.
  For Core Binding Factor (CBF) leukemia patients: Cytarabine 3000 mg/m2 IV twice daily (BID), 12 hours apart x 6 doses either on Days 1, 3, and 5 OR Days 1, 2, and 3 (per institutional preference) followed by Venetoclax 100 mg daily Day 1 through Day 8
  For non-Core Binding Factor (CBF) leukemia patients: Cytarabine 1500 mg/m2 IV twice daily (BID), 12 hours apart x 6 either on Days 1, 3, and 5 OR Days 1, 2, and 3 (per institutional preference) followed by Venetoclax 100 mg daily Day 1 through Day 8
  Interventions: Drug: Cytarabine; Drug: Venetoclax
- Arm C: Daunorubicin + Cytarabine Liposome+ Venetoclax (Experimental): Patients will participate for 2 cycles. Each cycle is 28 days.
  Daunorubicin 29 mg/m2/Cytarabine 65 mg/m2 liposome IV on Days 1 and 3 with Venetoclax 400 mg orally once daily on Days 1-14
  Interventions: Drug: Venetoclax; Drug: CPX-351
- Arm D: Azacitidine + Venetoclax (Experimental): Patients will participate for 2 cycles. Each cycle is 28 days.
  Azacitidine 75 mg/m2 IV/SC on Days 1-7 OR Days 1-5 and Days 8-9 (per institutional preference) with Venetoclax 400 mg orally once daily on Days 1-28
  Interventions: Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Cytarabine — Arm A: CBF-Cytarabine 3000 mg/m2 or 1500 mg/m2 IV twice daily (BID), 12 hours apart x 6 doses either on Days 1, 3, and 5 OR Days 1, 2, and 3
  Other Names: 63878
  Arms: Arm A: Cytarabine; Arm B: Cytarabine + Venetoclax
Drug: Venetoclax — Venetoclax 100 mg daily Day 1 through Day 8 Venetoclax 400 mg orally once daily on Days 1-14 Venetoclax 400 mg orally once daily on Days 1-28
  Other Names: Venclexta; 766270
  Arms: Arm B: Cytarabine + Venetoclax; Arm C: Daunorubicin + Cytarabine Liposome+ Venetoclax; Arm D: Azacitidine + Venetoclax
Drug: CPX-351 — Daunorubicin 29 mg/m2/Cytarabine 65 mg/m2 liposome IV on Days 1 and 3
  Other Names: Daunorubicin + Cytarabine Liposome; Vyxeos; 775341
  Arms: Arm C: Daunorubicin + Cytarabine Liposome+ Venetoclax
Drug: Azacitidine — Azacitidine 75 mg/m2 IV/SC on Days 1-7 OR Days 1-5 and Days 8-9 (per institutional preference)
  Other Names: Onureg; Vidaza; 102816
  Arms: Arm D: Azacitidine + Venetoclax

SUMMARY:
ERASE is part of the MyeloMATCH initiative, Young Adult Basket and is a Tier 2 study. The study is comparing the use of Cytarabine to Cytarabine and Venetoclax, Daunorubicin/Cytarabine Liposome and Venetoclax, and Azacitidine and Venetoclax.

DETAILED DESCRIPTION:
MM2YA-EA01 is a randomized Phase 2 study. Patients will be randomized to 1 of 4 treatment arms in a 1:1:1:1 ratio. The 4 treatment arms will compare: Cytarabine 3000 mg/m2 for CBD patients/1500 mg/m2 for non-CBD patients to cytarabine 3000 mg/m2 for CBD patients/1500 mg/m2 for non-CBD patients plus venetoclax 100 mg, daunorubicin 29 mg/m2/Cytarabine 65 mg/m2 liposome plus venetoclax 400 mg, and Azacitidine 75 mg/m2 plus venetoclax 400 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18 and ≤ 59 years of age.
* Patient must have ECOG performance status 0-2
* Patient must have morphologically documented AML or secondary AML [from prior conditions such as myelodysplastic syndrome (MDS), myeloproliferative neoplasm (MPN)] or therapy related AML (t-AML), as defined by World Health Organization (WHO) criteria
* Patient must have completed induction chemotherapy in a myeloMATCH Young Adult Tier-1 protocol. Patient may have received prior hypomethylating agents (HMAs). Patient may have received prior azacitidine + venetoclax.
* Patient must have been assigned to this protocol by myeloMATCH MSRP/MATCHBOX/. Patients thereby assigned will have attained complete remission (CR) or CR with partial hematologic recovery (CRh) (defined as CR with (ANC) ≥ 500/mcL and/or platelets > 50/mcL) with detectable MRD at time of assignment. MRD is defined as >0.1% flow cytometry on bone marrow (BM) biopsy as assessed by MDNet. The definition of CR or CRh may be made ± 2 weeks from BM biopsy
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.
* Patient must have recovered (i.e.: resolved to < grade 2) from adverse events related to prior anti-cancer therapy at the time of randomization with the exception of alopecia
* Patient must have adequate organ and marrow function as defined below (these labs must be obtained ≤ 7 days prior to protocol randomization):

Absolute neutrophil count (ANC) ≥ 500/mcL ANC:__________ Date of Test:__________ Platelets ≥ 50,000/mcL Platelets:__________ Date of Test:__________ Total bilirubin ≤ 2 x institutional upper limit of normal (ULN) Total Bilirubin:__________ Institutional ULN:_________ Date of Test:__________ AST(SGOT)/ALT(SGPT) ≤ 3.0 × institutional ULN AST:_______ Institutional ULN:_________ Date of Test:_______ ALT: _______Institutional ULN:_________ Creatinine ≤ 1.5 x institutional ULN Creatinine ______________Date of Test:________ OR

≥ 50 mL/min/1.73 m2

* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients must be able to swallow oral tablets and be free of GI absorption issues.

Exclusion Criteria:

* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.

All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy.

A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Patient of child bearing potential? ______ (Yes or No) Date of blood test or urine study: ___________

* Patients of childbearing potential and/or sexually active patients must not expect to conceive or father children by using an accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and continue for 6 months after the last dose of daunorubicin + cytrarabine liposome, 6 months after the last dose of azacitidine for patients of childbearing potential, 3 months after the last dose of azacitidine for male patients, and for 30 days after the last dose of venetoclax. Patient must also abstain from nursing an infant for 2 weeks after the last dose of daunorubicin + cytrarabine liposome and for 1 week after the last dose of azacitidine.
* Patients must not have FLT3 TKD or ITD mutation. Patients with this mutation, will be excluded from this study because myeloMATCH plans separate studies in tier-2 for those patients
* Patient must not be receiving any other investigational agents at the time of randomization.
* Patient must not have history of allergic reactions attributed to compounds of similar chemical or biologic composition to cytarabine, azacitidine, venetoclax or Daunorubicin and Cytarabine liposome
* Patients must not have uncontrolled intercurrent illness including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or serious chronic gastrointestinal conditions associated with diarrhea

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-10-23 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Rate of Achieving Minimal residual disease (MRD) | Day 56
  Rate of Achieving MRD Negative CR

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Atallah, MD, Study Chair — Medical College of Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araki D, Wood BL, Othus M, Radich JP, Halpern AB, Zhou Y, Mielcarek M, Estey EH, Appelbaum FR, Walter RB. Allogeneic Hematopoietic Cell Transplantation for Acute Myeloid Leukemia: Time to Move Toward a Minimal Residual Disease-Based Definition of Complete Remission? J Clin Oncol. 2016 Feb 1;34(4):329-36. doi: 10.1200/JCO.2015.63.3826. Epub 2015 Dec 14. PMID 26668349
- [Background] Othus M, Wood BL, Stirewalt DL, Estey EH, Petersdorf SH, Appelbaum FR, Erba HP, Walter RB. Effect of measurable ('minimal') residual disease (MRD) information on prediction of relapse and survival in adult acute myeloid leukemia. Leukemia. 2016 Oct;30(10):2080-2083. doi: 10.1038/leu.2016.120. Epub 2016 May 2. No abstract available. PMID 27133827
- [Background] Freeman SD, Hills RK, Virgo P, Khan N, Couzens S, Dillon R, Gilkes A, Upton L, Nielsen OJ, Cavenagh JD, Jones G, Khwaja A, Cahalin P, Thomas I, Grimwade D, Burnett AK, Russell NH. Measurable Residual Disease at Induction Redefines Partial Response in Acute Myeloid Leukemia and Stratifies Outcomes in Patients at Standard Risk Without NPM1 Mutations. J Clin Oncol. 2018 May 20;36(15):1486-1497. doi: 10.1200/JCO.2017.76.3425. Epub 2018 Mar 30. PMID 29601212
- [Background] Buccisano F, Maurillo L, Gattei V, Del Poeta G, Del Principe MI, Cox MC, Panetta P, Consalvo MI, Mazzone C, Neri B, Ottaviani L, Fraboni D, Tamburini A, Lo-Coco F, Amadori S, Venditti A. The kinetics of reduction of minimal residual disease impacts on duration of response and survival of patients with acute myeloid leukemia. Leukemia. 2006 Oct;20(10):1783-9. doi: 10.1038/sj.leu.2404313. Epub 2006 Jul 13. PMID 16838027
- [Background] Freeman SD, Virgo P, Couzens S, Grimwade D, Russell N, Hills RK, Burnett AK. Prognostic relevance of treatment response measured by flow cytometric residual disease detection in older patients with acute myeloid leukemia. J Clin Oncol. 2013 Nov 10;31(32):4123-31. doi: 10.1200/JCO.2013.49.1753. Epub 2013 Sep 23. PMID 24062403
- [Background] Terwijn M, van Putten WL, Kelder A, van der Velden VH, Brooimans RA, Pabst T, Maertens J, Boeckx N, de Greef GE, Valk PJ, Preijers FW, Huijgens PC, Drager AM, Schanz U, Jongen-Lavrecic M, Biemond BJ, Passweg JR, van Gelder M, Wijermans P, Graux C, Bargetzi M, Legdeur MC, Kuball J, de Weerdt O, Chalandon Y, Hess U, Verdonck LF, Gratama JW, Oussoren YJ, Scholten WJ, Slomp J, Snel AN, Vekemans MC, Lowenberg B, Ossenkoppele GJ, Schuurhuis GJ. High prognostic impact of flow cytometric minimal residual disease detection in acute myeloid leukemia: data from the HOVON/SAKK AML 42A study. J Clin Oncol. 2013 Nov 1;31(31):3889-97. doi: 10.1200/JCO.2012.45.9628. Epub 2013 Sep 23. PMID 24062400
- [Background] Pan R, Hogdal LJ, Benito JM, Bucci D, Han L, Borthakur G, Cortes J, DeAngelo DJ, Debose L, Mu H, Dohner H, Gaidzik VI, Galinsky I, Golfman LS, Haferlach T, Harutyunyan KG, Hu J, Leverson JD, Marcucci G, Muschen M, Newman R, Park E, Ruvolo PP, Ruvolo V, Ryan J, Schindela S, Zweidler-McKay P, Stone RM, Kantarjian H, Andreeff M, Konopleva M, Letai AG. Selective BCL-2 inhibition by ABT-199 causes on-target cell death in acute myeloid leukemia. Cancer Discov. 2014 Mar;4(3):362-75. doi: 10.1158/2159-8290.CD-13-0609. Epub 2013 Dec 17. PMID 24346116
- [Background] DiNardo CD, Lachowiez CA, Takahashi K, Loghavi S, Xiao L, Kadia T, Daver N, Adeoti M, Short NJ, Sasaki K, Wang S, Borthakur G, Issa G, Maiti A, Alvarado Y, Pemmaraju N, Montalban Bravo G, Masarova L, Yilmaz M, Jain N, Andreeff M, Jabbour E, Garcia-Manero G, Kornblau S, Ravandi F, Konopleva MY, Kantarjian HM. Venetoclax Combined With FLAG-IDA Induction and Consolidation in Newly Diagnosed and Relapsed or Refractory Acute Myeloid Leukemia. J Clin Oncol. 2021 Sep 1;39(25):2768-2778. doi: 10.1200/JCO.20.03736. Epub 2021 May 27. PMID 34043428
- [Background] Kadia TM, Reville PK, Borthakur G, Yilmaz M, Kornblau S, Alvarado Y, Dinardo CD, Daver N, Jain N, Pemmaraju N, Short N, Wang SA, Tidwell RSS, Islam R, Konopleva M, Garcia-Manero G, Ravandi F, Kantarjian HM. Venetoclax plus intensive chemotherapy with cladribine, idarubicin, and cytarabine in patients with newly diagnosed acute myeloid leukaemia or high-risk myelodysplastic syndrome: a cohort from a single-centre, single-arm, phase 2 trial. Lancet Haematol. 2021 Aug;8(8):e552-e561. doi: 10.1016/S2352-3026(21)00192-7. PMID 34329576
- [Background] Maiti A, DiNardo CD, Qiao W, Kadia TM, Jabbour EJ, Rausch CR, Daver NG, Short NJ, Borthakur G, Pemmaraju N, Yilmaz M, Alvarado Y, Montalbano KS, Wade A, Maduike RE, Guerrero JA, Vaughan K, Bivins CA, Pierce S, Ning J, Ravandi F, Kantarjian HM, Konopleva MY. Ten-day decitabine with venetoclax versus intensive chemotherapy in relapsed or refractory acute myeloid leukemia: A propensity score-matched analysis. Cancer. 2021 Nov 15;127(22):4213-4220. doi: 10.1002/cncr.33814. Epub 2021 Aug 3. PMID 34343352
- [Background] DiNardo CD, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Wei AH, Konopleva M, Dohner H, Letai A, Fenaux P, Koller E, Havelange V, Leber B, Esteve J, Wang J, Pejsa V, Hajek R, Porkka K, Illes A, Lavie D, Lemoli RM, Yamamoto K, Yoon SS, Jang JH, Yeh SP, Turgut M, Hong WJ, Zhou Y, Potluri J, Pratz KW. Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia. N Engl J Med. 2020 Aug 13;383(7):617-629. doi: 10.1056/NEJMoa2012971. PMID 32786187
- [Background] Cortes JE, Goldberg SL, Feldman EJ, Rizzeri DA, Hogge DE, Larson M, Pigneux A, Recher C, Schiller G, Warzocha K, Kantarjian H, Louie AC, Kolitz JE. Phase II, multicenter, randomized trial of CPX-351 (cytarabine:daunorubicin) liposome injection versus intensive salvage therapy in adults with first relapse AML. Cancer. 2015 Jan 15;121(2):234-42. doi: 10.1002/cncr.28974. Epub 2014 Sep 15. PMID 25223583
- [Background] Plesa A, Roumier C, Gutrin J, Larcher MV, Balsat M, Cadassou O, Barraco F, Fossard G, Baudouin A, Labussiere H, Tigaud I, Ducastelle S, Hayette S, Sujobert P, Heiblig M, Elhamri M, Thomas X. Measurable residual disease including AML leukemia stem cell flow evaluation of CPX-351 therapy by multi-parameter flow cytometry. Leuk Res. 2021 Dec;111:106673. doi: 10.1016/j.leukres.2021.106673. Epub 2021 Jul 26. No abstract available. PMID 34364023
- [Background] Kolitz JE, Strickland SA, Cortes JE, Hogge D, Lancet JE, Goldberg SL, Villa KF, Ryan RJ, Chiarella M, Louie AC, Ritchie EK, Stuart RK. Consolidation outcomes in CPX-351 versus cytarabine/daunorubicin-treated older patients with high-risk/secondary acute myeloid leukemia. Leuk Lymphoma. 2020 Mar;61(3):631-640. doi: 10.1080/10428194.2019.1688320. Epub 2019 Nov 25. PMID 31760835
- [Background] Mayer RJ, Davis RB, Schiffer CA, Berg DT, Powell BL, Schulman P, Omura GA, Moore JO, McIntyre OR, Frei E 3rd. Intensive postremission chemotherapy in adults with acute myeloid leukemia. Cancer and Leukemia Group B. N Engl J Med. 1994 Oct 6;331(14):896-903. doi: 10.1056/NEJM199410063311402. PMID 8078551
- [Background] Johnson-Farley N, Veliz J, Bhagavathi S, Bertino JR. ABT-199, a BH3 mimetic that specifically targets Bcl-2, enhances the antitumor activity of chemotherapy, bortezomib and JQ1 in "double hit" lymphoma cells. Leuk Lymphoma. 2015 Jul;56(7):2146-52. doi: 10.3109/10428194.2014.981172. Epub 2015 Jan 28. PMID 25373508
- [Background] Niu X, Zhao J, Ma J, Xie C, Edwards H, Wang G, Caldwell JT, Xiang S, Zhang X, Chu R, Wang ZJ, Lin H, Taub JW, Ge Y. Binding of Released Bim to Mcl-1 is a Mechanism of Intrinsic Resistance to ABT-199 which can be Overcome by Combination with Daunorubicin or Cytarabine in AML Cells. Clin Cancer Res. 2016 Sep 1;22(17):4440-51. doi: 10.1158/1078-0432.CCR-15-3057. Epub 2016 Apr 21. PMID 27103402
- [Background] Richard M. Stone, Daniel J. DeAngelo, Ilene Galinsky, Caroline Kokulis, Jeremy M. Stewart, Michael McGinnis, Lillian Werner, Anthony G. Letai, Marina Y Konopleva, Marlise Luskin; Phase I Trial of Escalating Doses of the Bcl-2 Inhibitor Venetoclax in Combination with Daunorubicin/Cytarabine Induction and High Dose Cytarabine Consolidation in Previously Untreated Adults with Acute Myeloid Leukemia ( AML). Blood 2019; 134 (Supplement_1): 3908. doi: https://doi.org/10.1182/blood-2019-124966
- [Background] Magina KN, Pregartner G, Zebisch A, Wolfler A, Neumeister P, Greinix HT, Berghold A, Sill H. Cytarabine dose in the consolidation treatment of AML: a systematic review and meta-analysis. Blood. 2017 Aug 17;130(7):946-948. doi: 10.1182/blood-2017-04-777722. Epub 2017 Jul 5. No abstract available. PMID 28679736
- [Background] Aldoss I, Yang D, Aribi A, Ali H, Sandhu K, Al Malki MM, Mei M, Salhotra A, Khaled S, Nakamura R, Snyder D, O'Donnell M, Stein AS, Forman SJ, Marcucci G, Pullarkat V. Efficacy of the combination of venetoclax and hypomethylating agents in relapsed/refractory acute myeloid leukemia. Haematologica. 2018 Sep;103(9):e404-e407. doi: 10.3324/haematol.2018.188094. Epub 2018 Mar 15. No abstract available. PMID 29545346
- [Background] Ganzel C, Ram R, Gural A, Wolach O, Gino-Moor S, Vainstein V, Nachmias B, Apel A, Koren-Michowitz M, Pasvolsky O, Yerushalmi R, Danylesko I, Cohen Y, Peretz G, Moshe Y, Zektser M, Yeganeh S, Rowe JM, Ofran Y. Venetoclax is safe and efficacious in relapsed/refractory AML. Leuk Lymphoma. 2020 Sep;61(9):2221-2225. doi: 10.1080/10428194.2020.1761964. Epub 2020 May 18. PMID 32420775
- [Background] Pratz KW, Jonas BA, Pullarkat V, Recher C, Schuh AC, Thirman MJ, Garcia JS, DiNardo CD, Vorobyev V, Fracchiolla NS, Yeh SP, Jang JH, Ozcan M, Yamamoto K, Illes A, Zhou Y, Dail M, Chyla B, Potluri J, Dohner H. Measurable Residual Disease Response and Prognosis in Treatment-Naive Acute Myeloid Leukemia With Venetoclax and Azacitidine. J Clin Oncol. 2022 Mar 10;40(8):855-865. doi: 10.1200/JCO.21.01546. Epub 2021 Dec 15. PMID 34910556